CLINICAL TRIAL: NCT07157540
Title: Testing the Effects of a Digital Intervention for Cannabis Harm Reduction - The Cann'App Fractional Factorial Randomized Controlled Trial
Brief Title: Testing the Effects of Cann'App, a Digital Intervention for Cannabis Harm Reduction
Acronym: Cann'App
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Jacques Gaume (Other)
Collaborators: Swiss National Science Foundation (Other); Apptitude (Unknown); Addiction Switzerland (Unknown)
Responsible Party: Sponsor-Investigator, Jacques Gaume, PhD scientist, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 2025-00428; 10001E_220072 (Other Grant/Funding Number: Swiss National Science Foundation)
Record Dates: First submitted 2025-08-27; First posted 2025-09-05 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Cannabis Use; Harm Reduction
Keywords: Protective Behavioral Strategies; Cannabis Use; Digital Intervention; Adult Regular Cannabis Users; Personalized Normative Feedback; Substance-Free Activity Session; Cannabis Harm Reduction; Counterfactual Thinking; Episodic Future Thinking; Web-Based Application; Cannabis Expenditures; Cannabis Related-Consequences
MeSH Terms: conditions — Harm Reduction

STUDY DESIGN:
Intervention Model Description: Monocentric 5-arm fractional factorial randomized controlled trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The randomization will be imbedded within the application, therefore concealment of allocation will be total. Participants will be blind to their experimental condition. Research staff involved in the study will not be informed of participants' group allocation. All study assessments will be done electronically. The generation of the randomization sequence and its programing into the study website will be conducted by the developing team who will not have contacts with participants or any involvement in the study implementation and analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Condition 1 - Personalized Feedback + Information (Experimental): Access to "Personalized Feedback" module (PF, Study Intervention) and "Information" module (Minimal, Control Intervention)
  Interventions: Behavioral: Personalized Feedback on Cannabis Protective Behavioral Strategies, Cannabis Use, Cannabis Expenditures, and Cannabis-Related Consequences (PF); Behavioral: Information
- Condition 2 - Imagine the future + Information (Experimental): Access to "Imagine the Future" module (IMAGIN, Study Intervention) and "Information" module (Minimal, Control Intervention)
  Interventions: Behavioral: Imagining the Future Using Counterfactual Thinking and Episodic Future Thinking (IMAGIN); Behavioral: Information
- Condition 3 - Substance-Free Activities Session + Information (Experimental): Access to "Substance-Free Activities Session" module (SFAS, Study Intervention) and "Information" module (Minimal, Control Intervention)
  Interventions: Behavioral: Behavioral Economics-Informed Exercises to Increase Motivation to Engage in Substance-Free Activities (SFAS); Behavioral: Information
- Condition 4 - Full Intervention + Information (Experimental): Access to the full intervention (PF+IMAGIN+SFAS) and "Information" module (Minimal, Control Intervention)
  Interventions: Behavioral: Personalized Feedback on Cannabis Protective Behavioral Strategies, Cannabis Use, Cannabis Expenditures, and Cannabis-Related Consequences (PF); Behavioral: Imagining the Future Using Counterfactual Thinking and Episodic Future Thinking (IMAGIN); Behavioral: Behavioral Economics-Informed Exercises to Increase Motivation to Engage in Substance-Free Activities (SFAS); Behavioral: Information
- Condition 5 - Information only (Control) (Active Comparator): Access to "Information" module (Minimal, Control Intervention)
  Interventions: Behavioral: Information

INTERVENTIONS:
Behavioral: Personalized Feedback on Cannabis Protective Behavioral Strategies, Cannabis Use, Cannabis Expenditures, and Cannabis-Related Consequences (PF) — PF comprises the following content:
  * Self-reported PBS questionnaire, personalized feedback on PBS, possibility to select strategies to start using or use more often, possibility to set a reminder to use PBS strategies.
  * Short questionnaire on cannabis use (frequency/number of hours under the influence) and normative feedback on participant's cannabis use as compared to people of same age and gender in the general population and among Cann-L participants.
  * Question on money spent for cannabis purchase, personalized feedback (total amount spent and corresponding number of grams of cannabis over one year), gamified gauge to picture potential yearly savings, reflection on how to use the saved money, and possibility to set a reminder for money saving objectives.
  * Questionnaire on cannabis-related consequences, feedback on the level of consequences met, question about which consequence(s) participant might want to think about, and possibility to set a reminder to think about consequences.
  Arms: Condition 1 - Personalized Feedback + Information; Condition 4 - Full Intervention + Information
Behavioral: Imagining the Future Using Counterfactual Thinking and Episodic Future Thinking (IMAGIN) — Two-task intervention including:
  1. Counterfactual thinking:
     * Description of a recent negative situation related to cannabis use encountered by the participant
     * Identification of a preventive strategy that would have addressed this situation
     * Writing a sentence formatted as "If only +preventive strategy, then + description on how the specific past problem would have improved"
     * Assessment of participant's intention and confidence in using the preventive strategy
     * Imagining a future situation using this preventive strategy
     * Possibility to set a reminder of the preventive strategy.
  2. Episodic future thinking:
     * Description of a significant positive event that might occur in the short-term (3 months) and that does not involve cannabis use
     * Assessment of the importance and enjoyment of this positive event
     * Encouragement to imagine it as vividly as possible
     * Suggestion to describe the positive event in detail and to write it down
     * Possibility to set a reminder of the positive event.
  Arms: Condition 2 - Imagine the future + Information; Condition 4 - Full Intervention + Information
Behavioral: Behavioral Economics-Informed Exercises to Increase Motivation to Engage in Substance-Free Activities (SFAS) — SFAS includes:
  * A questionnaire on how participant value different aspects of their life, and feedback on valued domains.
  * Two open-ended questions on short- and long-term life goals.
  * A questionnaire assessing time allocation (hours per week allocated to different activities, e.g. socializing, working, etc.), and personalized feedback including the time spent using substances and recovering from their effects.
  * Gamified exercise to imagine allocating time in a different way.
  * List of substance-free recreational activities in the region of Lausanne, with possibility to select activities on a "wish-list" including internet hyperlinks.
  * Possibility to set a reminder of the selected activities.
  * Single-item questionnaire on stress and mood, and feedback on stress and mood level.
  * Open-ended question on coping strategies currently used for stress and mood.
  * List of coping strategies that can be selected.
  * Possibility to set a reminder of stress/mood coping strategies.
  Arms: Condition 3 - Substance-Free Activities Session + Information; Condition 4 - Full Intervention + Information
Behavioral: Information — Minimal intervention (Control Intervention), consisting of simple, text-only web pages containing information on cannabis effects and health-related risks, cannabis consumption modes, cannabis harm reduction and protective behavioral strategies, as well as hyperlinks to additional resources and online help.

SUMMARY:
The goal of this clinical trial is to learn if a digital web application can prevent the risks related to cannabis use among adult regular cannabis users who are enrolled in a pilot trial for cannabis sales regulation conducted in Lausanne, Switzerland (i.e., Cann-L study) and have agreed that their data were used in other studies.

The main question it aims to answer is:

Do participants who have access to the intervention modules of the web application raise their use of protective behavioral strategies to lower cannabis-related risks?

Researchers will compare the intervention modules to a control module (i.e., information on cannabis-related risks and harm reduction) to see if the web application works to prevent the risks related to cannabis use. They will also compare intervention modules across each other to see whether one works better than another.

Participants will:

* Create a user account in the web application
* Access the web application using a laptop, tablet or smartphone
* Use the web application as they wish throughout the duration of the study
* Complete the regular Cann-L study questionnaires every six months, which will be used to measure their cannabis use and related risks.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will be those included in the pilot trial of cannabis sales regulation in Lausanne, Switzerland (Cann-L study).

Inclusion criteria in Cann-L study are:

* being adult (>18 years old),
* having current cannabis use (i.e., use at least once a month over the last 6 months)
* living in the city of Lausanne. To enter the study, they complete an entry assessment verifying their age and proof of residence, and confirming that they have current cannabis use.

Exclusion Criteria:

* Cann-L exclusion criteria comprise:
* being younger than 18 years old,
* being pregnant or breastfeeding,
* having a health condition contraindicating the use of cannabis (e.g., severe psychiatric disorder).

The consent to participate in the Cann-L parent trial comprises an option to be contacted to participate in sub-studies, including studies on prevention measures. All participants having accepted to be so contacted will be proposed to participate in the present study.

Therefore, additional exclusion criteria for the present study include:

* not providing informed consent to participate in sub-studies, including studies on prevention measures,
* not providing informed consent to participate in the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 565 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Frequency of Protective Behavioral Strategies for Marijuana Use as Measured by the PBSM-17 Short Form Scale | This outcome will be assessed at 1- and 7-month follow-up.
  This outcome will be measured using the Protective Behavioral Strategies for Marijuana Use (PBSM-17) Short Form scale, a self-reported 17-item questionnaire measuring the frequency of PBS for cannabis use on a 6-point Likert scale ranging from 1 (never) to 6 (always).

SECONDARY OUTCOMES:
Cannabis Use Frequency | This outcome will be measured at 1- and 7-month follow-up.
  Cannabis Use Frequency will be measured using a single item asking "During the past 30 days, on how many days did you use cannabis?"
Number of Hours High on a Typical Day | This outcome will be measured at 1- and 7-month follow-up.
  The number of hours under influence will be measured using a single item asking "How many total hours were you high on a typical day when you had been using cannabis?"

OTHER OUTCOMES:
Cannabis Use Disorder Severity as Measured by CUDIT-R | This outcome will be measured at 1- and 7-month follow-up.
  This outcome will be measured using the Cannabis Use Disorder Identification Test - Revised (CUDIT-R), a self-reported 8-items questionnaire (i.e., question 1-7 are scored on a 0-4 scale, and question 8 is scored 0, 2, or 4). Scores of 8 or more indicate hazardous cannabis use, while scores of 12 or more indicate a possible cannabis use disorder for which further intervention may be required.
Cannabis Purchase Task | This outcome will be assessed at 1- and 7-month follow-up.
  This outcome will be used to measure behavioral economics indices of cannabis demand. Participants will be asked to report hypothetical cannabis consumption in a scenario at escalating prices.
Source of Cannabis Supply | This outcome will be assessed at 1- and 7-month follow-up.
  This outcome will be measured for each cannabis product (herbal/marijuana, resin/hashish, oral oil, e-liquids, concentrates, edibles, other) by reporting the frequency of supply in a) Cann-L study dispensary, b) other external sources (e.g., acquaintances, on the street, social networks, darknet).
Alternatives to Smoking Cannabis | This outcome will be assessed at 1- and 7-month follow-up.
  The frequency of use of four main consumption modes (smoking, vaping/dabbing, absorbing, and edibles) will be measured using four corresponding cursors for which the total should be 100%.
Purchase of Cannabis with Lower THC Ratio | This outcome will be assessed at 1- and 7-month follow-up.
  This outcome will be computed based on individual sales data from Cann-L study dispensary.
Simultaneous Use of Cannabis and Other Substances | This outcome will be assessed at 1- and 7-month follow-up.
  This outcome will be assessed by two items measuring the frequency of simultaneous use, one for alcohol and one for other illegal drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Gaume, PhD, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- Lausanne University Hospital, Lausanne, Vaud Canton, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The data collected for this study may be reused and/or transmitted for other studies (including abroad), always in coded form (i.e., deidentified dataset). For each instance of reuse in another study, a data transfer agreement will need to be established.
Time Frame: Beginning immediately after the publication of results and ending 20 years after study termination.
Access Criteria: A formal request should be submitted to the Principal investigator and a data sharing agreement must be signed.